CLINICAL TRIAL: NCT05157659
Title: A Clinical Imaging Study Using [18F]F-AraG PET to Visualize Tumor Infiltrating T-cell Activation in Non-small Cell Lung Cancer.
Brief Title: [18F]F-AraG PET Imaging to Visualize Tumor Infiltrating T-cell Activation in Non-small Cell Lung Cancer.
Acronym: ATTAIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Idris Bahce, dr. I. Bahce, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL77310.029.21; 2021-001489-40 (EudraCT Number)
Record Dates: First submitted 2021-12-01; First posted 2021-12-15 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Positron Emission Tomography; [18F]F-AraG; T-Lymphocytes; Kinetic Modelling; Reproducibility of Results
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]F-AraG PET procedures (Experimental): Within one week prior to resection two [18F]F-AraG PET-scans will be performed.
  Interventions: Diagnostic Test: [18F]F-AraG PET-scan

INTERVENTIONS:
Diagnostic Test: [18F]F-AraG PET-scan — [18F]F-AraG PET scans are performed to assess the accumulation of activated T-cells in the tumour and healthy tissue.

SUMMARY:
[18F]F-AraG is a promising tracer to image activated T-cells with positron emission tomography (PET). The aim of the ATTAIN trial is to investigate the pharmacokinetic characteristics of this novel tracer by performing a full kinetic modelling, assess test-retest (TRT) variability and to correlate the tumor tracer uptake with the pathological assessment.

DETAILED DESCRIPTION:
The efficacy of immunotherapy and patient selection for combinatorial immunotherapy strategies would greatly improve if the tumor microenvironment (TME) could be characterized more accurately. Positron emission tomography (PET) using tracers that target immune cell subsets may provide a non-invasive means to immune profile the TME. Imaging T-cells can help in identifying 'hot' tumors, or parts of the tumor mass that have high concentrations of tumor infiltrating T-cells and also provide information on its activation.

A promising tracer to image activated T-cells is [18F]F-AraG. Based on the hypothesis that [18F]F-AraG will accumulate in activated T-cells, it is expected that [18F]F-AraG and PET will enable to (reproducibly) identify tumors and tumor areas with high concentrations of tumor infiltrating activated T-cells on pathological assessment. In the ATTAIN trial this [18F]F-AraG uptake in tumor lesions and healthy organs is explored by full kinetic modelling.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed NSCLC, a histological biopsy is mandatory.
2. Patients that are resectable upfront as per multidisciplinary tumor board evaluation.
3. Be willing and able to provide written informed consent for the trial.
4. Be above 18 years of age on day of signing informed consent.
5. Have a performance status of 0-1 on the ECOG Performance Scale at screening.

Exclusion Criteria:

1. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of screening. Inhaled or topical steroids, and adrenal replacement steroid >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
2. Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
3. Patient is pregnant or breastfeeding or expecting to conceive within the projected duration of the trial, starting with the screening visit through 12 weeks after the last [18F]F-AraG PET scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Full kinetic modelling | six months
  To perform full kinetic modeling of [18F]F-AraG for the uptake in tumor lesions and healthy organs (e.g. spleen) by exploring different kinetic models and outcome measures as well as its test-retest (TRT) variability to guide the selection of an optimal PET pharmacokinetic model.
Correlation with number of CD8 T-cell | six months
  To correlate the relationship between the tumor uptake of [18F]F-AraG and the number of CD8 T-cells amongst others as measured by Immunohistochemistry (IHC) and gene expression.

SECONDARY OUTCOMES:
Correlation with [18F]-FDG PET uptake | six months
  To correlate the [18F]-FDG PET uptake with uptake derived from [18F]F-AraG PET

OTHER OUTCOMES:
Correlation with immune profile of PBMCs | one year
  To explore the [18F]F-AraG PET uptake in tumor, lymph nodes and spleen with the immune profile of peripheral blood mononuclear cells (PBMC).

CONTACTS AND LOCATIONS:
Overall Officials: I. Bahce, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VU University Medical Center, Amsterdam, Nederland, Netherlands